CLINICAL TRIAL: NCT07063641
Title: Development of a Predictive Model to Identify Clinical Factors Associated With Response to Percutaneous Electrical Nerve Stimulation in Patients With Subacromial Pain Syndrome
Brief Title: Predictive Model for PENS Response in Subacromial Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Néstor Requejo Salinas (Other)
Collaborators: University of Alcala (Other); Centro Universitario La Salle (Other)
Responsible Party: Sponsor-Investigator, Néstor Requejo Salinas, Principal Investigator, Department of Physiotherapy, University of Alcalá and Centro Superior Universitario La Salle, Centro Universitario La Salle
Organization: Centro Universitario La Salle (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PENS-SDS-UAH-2025
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Subacromial Pain Syndrome; Rotator Cuff Related Shoulder Pain
Keywords: Percutaneous Electrical Nerve Stimulation; Suprascapular Nerve; Neural Mechanosensitivity; Musculoskeletal Pain; Ultrasound-Guided Interventions; Subacromial pain syndrome
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Uncontrolled, single-arm clinical trial aimed at developing a multivariable predictive model of response to suprascapular nerve-targeted PENS in patients with subacromial pain syndrome.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suprascapular Nerve PENS (Experimental): Participants in this arm will receive a single ultrasound-guided session of percutaneous electrical nerve stimulation (PENS) targeting the suprascapular nerve. The procedure involves needle placement adjacent to the suprascapular nerve and electrical stimulation for 30 minutes.
  Interventions: Device: Percutaneous Electrical Nerve Stimulation (PENS)

INTERVENTIONS:
Device: Percutaneous Electrical Nerve Stimulation (PENS) — Ultrasound-guided percutaneous electrical nerve stimulation applied to the suprascapular nerve using a monophasic or biphasic current at 10 Hz frequency and 250 μs pulse width. Intensity is progressively increased to patient tolerance, aiming to induce visible muscle contractions of the supraspinatus and infraspinatus. Duration of the session is 30 minutes.

SUMMARY:
Subacromial pain syndrome (SPS) is one of the most common causes of shoulder pain, leading to significant disability and socioeconomic burden. Although percutaneous electrical nerve stimulation (PENS) targeting the suprascapular nerve (SN) has shown positive therapeutic outcomes, individual response to the intervention varies considerably. This study aims to develop a multivariable predictive model to estimate clinical response to SN-targeted PENS in patients with SPS. The model will be built using clinical, psychological, and neural mechanosensitivity variables. The goal is to enhance patient selection and guide personalized treatment strategies.

DETAILED DESCRIPTION:
Subacromial pain syndrome (SPS) includes a group of clinical entities related to rotator cuff tendinopathy and subacromial structures that cause shoulder pain and functional limitations. PENS applied to the suprascapular nerve (SN) has demonstrated effectiveness in reducing pain and improving short-term function in patients with SPS. However, variability in clinical response suggests the influence of individual characteristics that are not yet well understood.

This study will conduct a prospective, single-arm, uncontrolled clinical trial involving 269 patients diagnosed with SPS. All participants will undergo a single ultrasound-guided session of PENS on the SN. The primary outcome will be post-treatment pain intensity measured with the Visual Analogue Scale (VAS). n addition to the primary outcome, several baseline variables will be collected to develop a multivariable beta regression predictive model. These variables include demographic data (age, sex, weight, height, BMI), clinical characteristics (pain duration in weeks, baseline pain intensity measured with the Visual Analogue Scale), psychological measures (Hospital Anxiety and Depression Scale - HADS), physical activity levels (International Physical Activity Questionnaire - Short Form), and measures of neural mechanosensitivity (pressure pain threshold on the infraspinatus and result of the suprascapular neurodynamic test). These predictors will be incorporated into the model regardless of their univariate significance, in line with best practices in predictive modelling.

A beta regression model will be developed to predict post-treatment pain intensity. Internal validation and model stability will be assessed using bootstrap resampling methods. This protocol follows the TRIPOD guidelines for clinical prediction model development.

Identifying reliable predictors of response will support clinical decision-making, helping to personalize physiotherapy approaches and improve the cost-effectiveness of SPS management. The findings may provide a robust foundation for future research and eventual clinical implementation of prediction tools for individualized therapy planning.

ELIGIBILITY:
Inclusion Criteria:

Adults aged between 18 and 65 years.

Clinical diagnosis of subacromial pain syndrome (SAPS), based on the following clinical criteria:

* Pain localized to the anterolateral shoulder region.
* Symptoms present for more than 6 weeks.
* Painful arc during shoulder abduction.
* Positive Neer or Hawkins-Kennedy impingement signs.
* Positive Jobe (empty can) test or external rotation resistance test.

Visual Analogue Scale (VAS) for shoulder pain ≥ 3/10 in the previous week.

Able to understand study procedures and sign informed consent.

Exclusion Criteria:

* Bilateral shoulder pain.
* History of fracture, dislocation, or surgical intervention on the affected shoulder.
* Presence of other shoulder pathologies such as adhesive capsulitis (frozen shoulder), glenohumeral instability, or full-thickness rotator cuff tear.
* Medical contraindications for PENS application (e.g., active anticoagulation, pregnancy, or decompensated psychiatric condition).
* Diagnosed cervical radiculopathy or myelopathy.
* Neurological or cognitive disorders interfering with study participation.
* Presence of chronic widespread pain syndromes, such as fibromyalgia.
* Belonephobia (severe needle phobia) that prevents intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks post-intervention
  Pain intensity will be measured with a 100 mm Visual Analogue Scale (VAS), ranging from 0 mm (no pain) to 100 mm (worst imaginable pain). This is the primary outcome used to evaluate the clinical response to a single ultrasound-guided session of percutaneous electrical nerve stimulation (PENS) targeting the suprascapular nerve in patients with subacromial pain syndrome. This outcome will be used as the dependent variable in the multivariable predictive model.

IPD SHARING:
Plan to Share IPD: Undecided